CLINICAL TRIAL: NCT01728168
Title: Prevalence of Food Allergies to Proteins From Different Legumes (Lupin, Peanut, Soy, and Pea) in Atopic and Healthy Subjects
Brief Title: Prevalence of Food Allergies to Proteins From Different Legumes
Status: Completed | Type: Observational
Sponsor: University of Jena (Other)
Collaborators: SRH Wald-Klinikum Gera GmbH (Other); German Federal Ministry of Education and Research (Other Government)
Responsible Party: Principal Investigator, Gerhard Jahreis, Prof. Dr. habil., University of Jena
Other Study IDs: LSEP H54-12
Record Dates: First submitted 2012-11-12; First posted 2012-11-16 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-02

CONDITIONS: Food Allergy
Keywords: lupin; peanut; soy; pea; legumes; cross-reactivity; sensitization; atopy
MeSH Terms: conditions — Food Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- Atopic: Subjects with either documented allergy, neurodermatitis, allergic asthma, allergic rhinitis, and/or a positive atopic score based on the criteria of Erlangen (>10 points).
- Non-atopic: Subjects without atopy.

SUMMARY:
The objective of the study is to assess the prevalence of a sensitization to proteins from legumes by skin prick test using commercial extracts (peanut, soy, and pea) and raw material (lupin) in atopic and healthy subjects.

ELIGIBILITY:
1. Inclusion Criteria:

   * Male and female subjects
   * Age 18 up to 75 years
   * For group "Atopic": either documented allergy, neurodermatitis, allergic asthma, allergic rhinitis, and/or a positive atopic score based on the criteria of Erlangen (>10 points).
2. Exclusion Criteria:

   * Intake of antihistamines, tricyclic antidepressants, systemic corticosteroids
   * Acute allergic symptoms
   * Skin infections at the test side
   * Pregnancy, lactation
   * Acute inflammatory diseases

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male and female subjects. Age: 18 to 75 years. Subjects with Atopy or non-atopic subjects.
Sampling Method: Non-Probability Sample
Enrollment: 183 (Actual)
Dates: Start 2012-12; Primary Completion 2013-07 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Evidence of a sensitization to legume proteins | 20 minutes after skin prick
  Evidence of a sensitization to one or more legume proteins (lupin, peanut, soy, and pea)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Kaatz, Dr. med., Study Director — SRH Wald-Klinikum Gera GmbH
Locations (1):
- SRH Wald-Klinikum Gera gGmbH, Gera, Thuringia, Germany